CLINICAL TRIAL: NCT07304973
Title: Vascular Endovascular Therapy: A Nurse-Led Predictive Nursing Protocol for Neurological Complications-Development, Validation, and Clinical Impact
Brief Title: Nurse-Led Predictive Protocol Cuts Neuro-Endovascular Complications
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Zhigang Lan, Professor, West China Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: WestChinaH-HX-2025-01
Record Dates: First submitted 2025-12-02; First posted 2025-12-26 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Endovascular Therapy; Neurological Complications
Keywords: Predictive nursing; Nurse-led checklist; Early intervention

STUDY DESIGN:
Intervention Model Description: Nurses used the predictive checklist to assess patients at 6 hours, 12 hours, 24 hours, and 48 hours postprocedural. For each assessment, items were scored as "positive" (1 point) or "negative" (0 point). A total score ≥4 points was defined as high risk, triggering immediate actions: (1) increased monitoring frequency (vital signs every 15 minutes, neurological assessment every 1 hour); (2) urgent cranial CT/MRI scan; (3) notification of the neurointerventional team within 10 minutes; (4) initiation of targeted interventions (e.g., blood pressure control, anti-edema therapy) as per protocol.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Nurses used the predictive checklist to assess patients at 6 hours, 12 hours, 24 hours, and 48 hours postprocedural. For each assessment, items were scored as "positive" (1 point) or "negative" (0 point). A total score ≥4 points was defined as high risk, triggering immediate actions: (1) increased monitoring frequency (vital signs every 15 minutes, neurological assessment every 1 hour); (2) urgent cranial CT/MRI scan; (3) notification of the neurointerventional team within 10 minutes; (4) initiation of targeted interventions (e.g., blood pressure control, anti-edema therapy) as per protocol.
  Interventions: Other: predictive checklist
- Control group (No Intervention): Patients received standard post-EVT care, including vital sign monitoring (every 15-30 minutes for the first 6 hours, then every 1-2 hours), neurological assessment (every 4 hours), and routine laboratory and imaging examinations (e.g., cranial CT at 24 hours postprocedural). Nurses documented clinical findings in electronic medical records and notified physicians only when obvious abnormalities were detected (e.g., NIHSS score increase ≥4 points, severe hypertension).

INTERVENTIONS:
Other: predictive checklist — Nurses used the predictive checklist to assess patients at 6 hours, 12 hours, 24 hours, and 48 hours postprocedural. For each assessment, items were scored as "positive" (1 point) or "negative" (0 point). A total score ≥4 points was defined as high risk, triggering immediate actions: (1) increased monitoring frequency (vital signs every 15 minutes, neurological assessment every 1 hour); (2) urgent cranial CT/MRI scan; (3) notification of the neurointerventional team within 10 minutes; (4) initiation of targeted interventions (e.g., blood pressure control, anti-edema therapy) as per protocol.
  Arms: Intervention Group

SUMMARY:
The goal of this prospective cohort study was to develop and test a 12-item, nurse-led predictive checklist that can quickly identify patients at high risk for neurological complications (bleeding, re-blockage, brain swelling, etc.) after endovascular therapy (EVT) for stroke or unruptured aneurysms. The main questions it aims to answer are:

Does the checklist accurately flag complications (sensitivity/specificity)? Does its use shorten the time between first abnormal sign and physician action? Does it lower the rate of severe complications or death and shorten hospital stay? Researchers compared 213 patients managed with the checklist (intervention group) to 213 patients who received standard nursing observation (control group).

Participants were:

Assessed by nurses at 6, 12, 24, and 48 hours post-EVT with the checklist (intervention) or usual monitoring (control) Followed for 7 days for any neurological complication and for 30 days for severe outcomes Checked with urgent CT/MRI and treated whenever the checklist score indicated high risk (≥4/12 points)

ELIGIBILITY:
Inclusion Criteria:

* 18 years old, underwent EVT for AIS (due to anterior circulation large vessel occlusion) or UIAs (size ≥5 mm)

  * had a postoperative stay of ≥48 hours.

Exclusion Criteria:

* preprocedural intracranial hemorrhage;
* severe liver or kidney dysfunction;
* coagulation disorders;
* refusal to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 426 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
AUC of the checklist | 7 days
  AUC of the checklist for predicting any neurological complication (HT, reocclusion, MCE, sICH) within 7 days postprocedural. Complications were diagnosed by neurointerventional physicians based on clinical manifestations and imaging findings (CT/MRI).

SECONDARY OUTCOMES:
incidence of severe complications | 30 days
  incidence of severe complications (defined as complications requiring surgical intervention, mechanical ventilation, or leading to death within 30 days);
length of hospital stay | 30 days
30-day mortality | 30 days

CONTACTS AND LOCATIONS:
Locations (1):
- West China Hospital, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: Yes
Protocol and informed consent